CLINICAL TRIAL: NCT05940220
Title: Efficacy of Oral Acetazolamide as Add-on Diuretic Therapy in Decongestion in Patients With Heart Failure and Diuretic Resistance
Brief Title: Efficacy of Oral Acetazolamide in Decongestion in Patients With Heart Failure
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IR.TUMS.THC.REC.1402.016
Record Dates: First submitted 2023-07-03; First posted 2023-07-11 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-06

CONDITIONS: Heart Failure
Keywords: : Acetazolamide, Heart failure, Electrolyte Disturbance, Diuretics, Chloride, Diuretic resistance, Decongestion
MeSH Terms: conditions — Heart Failure | interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- acetazolamid (Active Comparator): We will administer injectable and oral furosemide in infusion ward based on the dosage determined by the specialist on day zero. After that, we continue oral furosemide administration for three days. The prescribed dose of injectable and oral furosemide is determined by the specialist based on previous visits and hospitalizations in such a way that the patient has the least symptoms. The intervention group will receive acetazolamide 500 mg on day zero, then 250 mg bd for two days and 250 mg on the third day. The control group will receive placebo equivalent to acetazolamide.
  Interventions: Other: Acetazolamide
- placebo (Placebo Comparator): Acetazolamide placebo add-on a standard therapy of iv furosemide in one day and oral furosemide during three consecutive days will be used for the comparator arm.
  Interventions: Other: placebo

INTERVENTIONS:
Other: Acetazolamide — Acetazolamide placebo add-on a standard therapy of iv furosemide in one day and oral furosemide during three consecutive days will be used for the comparator arm
  Arms: acetazolamid
Other: placebo — placebo
  Arms: placebo

SUMMARY:
This is a 1:1 ratio single-center, double-blind, randomized controlled trial, aiming to enroll 130 patients admitted in infusion ward. The participants receive furosemide as standard treatment and will randomize towards 250 mg oral acetazolamide twice a day versus placebo on three consecutive days. The main objective is to determine the effect of oral acetazolamide and furosemide combination therapy on the decongestion. Prespecified secondary objectives included N-terminal pro B-type natriuretic peptide level on the 30th day, the readmission rate in a three-month period, quality of life assessment by Heart Failure Quality of Life Questionnaire at the end of the third month, change in weight, creatinine level, urinary sodium excretion, potassium level, and hematological indices in complete blood count at third day of the trial.

DETAILED DESCRIPTION:
This is a 1:1 ratio single center, double-blind, RCT on the diuretic and decongestive effects of oral acetazolamide in Iranian patients with HF. This study will be conducted on heart failure patients whose symptoms of congestion are not relieved by oral diuretics and are temporarily hospitalized in a section called the infusion ward and receive intravenous diuretics. The infusion unit is a separate unit where patients with heart failure who are not adequately relieved by oral diuretics are admitted for a short period of time and receive injectable furosemide. In this study, 250 mg acetazolamide tablets and placebo and furosemide 20 mg will be used. The medical information of the patients will be recorded, patients' clinical status will be evaluated by calculating the EVEREST score at baseline and third day , the weight and laboratory indices will also be measured at baseline and third day based on the same scale and fixed laboratory kits, respectively. Blood pressure will be also measured by an expert nurse at the baseline and each day before the furosemide injection by the same blood pressure cuff. Patients will be followed for clinical events to day 90. The protocol was drafted according to the standard protocol items for clinical trials) SPIRIT) guideline for randomized clinical trial protocols.

Study objectives The main objective is to determine the effect of oral acetazolamide and furosemide, as a loop diuretic, combination therapy on improvement of the congestion in patients at baseline and third day. Urinary sodium to creatinine ratio is an indicator in this objective and will be measured at 2 P.M. in these days.

Prespecified secondary objectives included the following: N-terminal pro B-type natriuretic peptide (NT-proBNP) level on the 30th day, the hospitalization rate in a three-month period, comparison of quality of life between two groups at the end of the third month and change in weight, creatinine level, urinary sodium excretion, potassium level, and hematological indices in complete blood count (CBC) at third day of the trial. At the end of the third month, we will assess our patients' quality of life using the Iranian Heart Failure Quality of Life (IHFQoL) Questionnaire. The validity and reliability of this questionnaire, which has 16 questions in 5 dimentions, has been confirmed by Naderi et al in 2012. (Kornbach's alpha coefficient= 0.922) .This questionnaire offers a range of total scores between 20 and 66. The items are scored on a three- or four-point Likert scale, with a higher score indicating a better quality of life for the individual. These are the five dimensions that are the subject of this survey: severity of disease symptoms (items 1, 2, 3, 4, 6), physical limitations (items 7-1 to 7-6), mental limitations (items 5, 9, 11), social aspects (items 8, 10, 12, 13), self-care (items 14, 15) and the patient's overall satisfaction (item 16). (16)

ELIGIBILITY:
Inclusion criteria

1. Earn at least 8 points from EVEREST score (see Table 1.)
2. Adult patients (≥ 18 years)
3. A major clinical sign of volume overload including edema, ascites confirmed by abdominal ultrasound, or pleural effusion confirmed by chest x-ray or chest ultrasound without using iv furosemide.
4. Maintenance treatment with oral furosemide as a loop diuretic ≥20 mg for at least one month
5. Using SGLT2i drugs including canagliflozin, dapagliflozin, and empagliflozin for at least one month

Exclusion criteria

1. Systolic blood pressure less than 90 mmHg or mean arterial pressure less than 65 mmHg
2. Estimated glomerular filtration rate (eGFR) <20 ml/min/1.73 m2
3. Using any diuretic agent except mineralocorticoid receptor antagonists including spironolactone and eplerenone
4. Simultaneous diagnosis of acute coronary syndrome, which is characterized by typical chest pain in addition to an increase in troponin level above the 99th percentile or electrocardiographic changes indicating ischemia or hospitalization as unstable angina.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-12-30 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Na/cr Ratio | baseline and third day
  . Urinary sodium to creatinine ratio is an indicator in this objective and will be measured at 2 P.M. in these days.

SECONDARY OUTCOMES:
N-terminal pro B-type natriuretic peptide (NT-proBNP) level | 30th day
  N-terminal pro B-type natriuretic peptide (NT-proBNP) level
Iranian Heart Failure Quality of Life (IHFQoL) Questionnaire | 3 months
  This questionnaire offers a range of total scores between 20 and 66

CONTACTS AND LOCATIONS:
Locations (1):
- Houshang bavandpour karvane, Tehran, Tehran Heart Center, Iran

IPD SHARING:
Plan to Share IPD: Undecided